CLINICAL TRIAL: NCT00316264
Title: A Phase 2, Randomized, Double-Blind Study to Evaluate the Safety, Tolerability, and Immunogenicity of Motavizumab (MEDI-524), a Humanized Enhanced Potency Monoclonal Antibody Against Respiratory Syncytial Virus (RSV), and Palivizumab When Administered in the Same Season
Brief Title: Study of Motavizumab (MEDI-524) and Palivizumab Administered Sequentially in the Same Respiratory Syncytial Virus (RSV) Season
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MI-CP127
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Results first posted 2012-12-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-11

CONDITIONS: Respiratory Syncytial Virus Infections; Chronic Lung Disease and <= 24 Months of Age or; Premature With Gestational Age <=35 Weeks and <=6 Months of Age
Keywords: Respiratory Syncytial Virus; Premature and under 6 mos. of age; Chronic Lung Disease over 6 mos. of age; palivizumab; motavizumab; RSV
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Premature Birth | interventions — motavizumab; Palivizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Motavizumab followed by Palivizumab (Experimental): 2 doses of motavizumab (15 mg/kg, administered as an intramuscular injection once/month) followed by 3 doses of palivizumab (15 mg/kg, administered as an intramuscular injection once/month)
  Interventions: Biological: Motavizumab, palivizumab
- Palivizumab followed by motavizumab (Experimental): 2 doses of palivizumab (15 mg/kg, administered as an intramuscular injection once/month) followed by 3 doses of motavizumab (15 mg/kg, administered as an intramuscular injection once/month)
  Interventions: Biological: Palivizumab, motavizumab
- Motavizumab control (Experimental): 5 doses of motavizumab (15 mg/kg, administered as an intramuscular injection once/month)
  Interventions: Biological: Motavizumab

INTERVENTIONS:
Biological: Motavizumab, palivizumab — Motavizumab was provided in sterile vials containing 100 mg of motavizumab in 1 mL of a sterile preservative-free liquid product at pH 6.0, formulated with 25 mM histidine-HCl.
  Arms: Motavizumab followed by Palivizumab
Biological: Palivizumab, motavizumab — Palivizumab was provided in sterile vials containing 100 mg of palivizumab in 1 mL of a sterile preservative-free liquid product at pH 6.0, formulated with 25 mM histidine, and 1.6 mM glycine.
  Arms: Palivizumab followed by motavizumab
Biological: Motavizumab — Motavizumab was provided in sterile vials containing 100 mg of motavizumab in 1 mL of a sterile preservative-free liquid product at pH 6.0, formulated with 25 mM histidine-HCl.
  Arms: Motavizumab control

SUMMARY:
This is a Phase 2, randomized, double-blind study in which motavizumab (MEDI-524) and palivizumab were administered sequentially to high-risk children during the same respiratory syncytial virus (RSV) season. A control group was administered only motavizumab.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind study in which motavizumab and palivizumab were administered sequentially to high-risk children during the same RSV season. It was anticipated that approximately 240 children (80 in each group) would be enrolled from the southern hemisphere during the upcoming RSV season (2006). Children were randomized into one of three regimens in a 1:1:1 ratio; the first group received 2 doses of motavizumab followed by 3 doses of palivizumab; the second group received 2 doses of palivizumab followed by 3 doses of motavizumab; and the third group received 5 doses of motavizumab. Motavizumab or palivizumab was administered at 15 mg/kg by IM injection every 30 days, for a total of 5 injections.

ELIGIBILITY:
Inclusion Criteria:

* The child must have been born at less than or equal to 35 weeks gestation and be less than or equal to 6 months of age at the time of entry into the study (child must be entered on or before his/her 6-month birthday); or the child must be less than or equal to 24 months of age at the time of entry into the study (child must be entered on or before his/her 24-month birthday) and diagnosed with chronic lung disease (CLD) of prematurity with stable or decreasing doses of diuretics, steroids, or bronchodilators, or treatment with supplemental oxygen, within the previous 6 months.
* The child must be in general good health at the time of study entry.
* The child's parent(s)/legal guardian must provide written informed consent.
* The child must be able to complete the follow-up visits through 120-150 days from last injection of study drug.
* Parent(s)/legal guardian of patient must have available telephone access.

Exclusion Criteria:

* Hospitalized at the time of study entry (unless discharge is expected within 10 days after entry into the study)
* Receiving chronic oxygen therapy or mechanical ventilation at the time of study entry (including continuous positive airway pressure [CPAP])
* Congenital heart disease (CHD) (children with medically or surgically corrected [closed] patent ductus arteriosus and no other CHD may be enrolled)
* Evidence of infection with hepatitis A, B, or C virus
* Known renal impairment, hepatic dysfunction, chronic seizure disorder, or immunodeficiency or HIV infection (a child of a mother with known HIV infection must be proven to be uninfected at the time of enrollment)
* Suspected serious allergic or immune-mediated events with prior receipt of palivizumab
* Acute illness or progressive clinical disorder
* Active infection, including acute RSV infection, at the time of enrollment
* Previous reaction to intravenous immunoglobulin (IGIV), blood products, or other foreign proteins
* Received within the past 120 days or currently receiving immunoglobulin products (such as RSV-IGIV [RespiGam], IVIG, or palivizumab) or any investigational agents
* Previous participation in a clinical trial of motavizumab
* Currently participating in any investigational study

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Actual)
Dates: Start 2006-04; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Griffin, M.D., Study Director — MedImmune LLC
Locations (19):
- Australia (7):
  - Department of Paediatrics and Child Health, The Canberra Hospital, Garran, Australian Capital Territory
  - Neonatalogy John Hunter Hospital, New Lambton Heights, New South Wales
  - Caboolture Clinical Research, Caboolture, Queensland
  - University of Queensland, Royal Children's Hospital, Herston, Queensland
  - Peninsula Clinical Research Centre, Kippa-Ring, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Respiratory Medicine Department, Royal Children's Hospital, Parkville, Victoria
- Chile (7):
  - Hospital Clinico de la Universidad de Chile, Independencia, Santiago Metropolitan
  - Hospital San Jose, Independencia, Santiago Metropolitan
  - Hospital Clinico de la Pontificia Universidad Catolica de Chile, Santiago
  - Hospital Clinico San Borja Arriaran, Santiago
  - Hospital Dr Felix Bulnes Cerda, Santiago
  - Hospital Dr. Sotero del Rio, Santiago
  - Hospital Padre Hurtado, Santiago
- New Zealand (5):
  - Kidz First, Middlemore Hospital, Otahuhu, Auckland
  - Christchurch Women's Hospital, Christchurch
  - Paediatric Medicine, Dunedin Hospital, Dunedin
  - Department of Paediatrics, Waikato Hospital, Hamilton
  - Child Health, Palmerston North Hospital, Palmerston North

REFERENCES:
- [Result] Fernandez P, Trenholme A, Abarca K, Griffin MP, Hultquist M, Harris B, Losonsky GA; Motavizumab Study Group. A phase 2, randomized, double-blind safety and pharmacokinetic assessment of respiratory syncytial virus (RSV) prophylaxis with motavizumab and palivizumab administered in the same season. BMC Pediatr. 2010 Jun 3;10:38. doi: 10.1186/1471-2431-10-38. PMID 20525274

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was anticipated that approximately 240 children (80 in each group) would be enrolled from the southern hemisphere during the upcoming RSV season (2006).
Pre-assignment Details: Children were randomized into one of three regimens in a 1:1:1 ratio; the first group received 2 doses of motavizumab followed by 3 doses of palivizumab; the second group received 2 doses of palivizumab followed by 3 doses of motavizumab; and the third group received 5 doses of motavizumab.
Groups:
- Motavizumab (MEDI-524) Followed by Palivizumab: 2 doses of motavizumab (15 mg/kg, administered as an intramuscular injection once/month) followed by 3 doses of palivizumab (15 mg/kg, administered as an intramuscular injection once/month)
- Palivizumab Followed by Motavizumab (MEDI-524): 2 doses of palivizumab (15 mg/kg, administered as an intramuscular injection once/month) followed by 3 doses of motavizumab (15 mg/kg, administered as an intramuscular injection once/month)
- Motavizumab (MEDI-524) Control: 5 doses of motavizumab (15 mg/kg, administered as an intramuscular injection once/month)
Period: Overall Study
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Started | 83 | 84 | 93
Completed | 77 | 77 | 87
Not Completed | 6 | 7 | 6
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal of Consent | 3 | 5 | 6
Not completed — Death | 2 | 0 | 0
Not completed — Other | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control | Total
Number analyzed (Participants) | 83 | 84 | 93 | 260
Age Continuous [Mean (Standard Deviation); unit: months] | 3.68 (3.13) | 3.35 (2.25) | 3.92 (2.43) | 3.66 (2.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 41 | 45 | 118
  Male | 51 | 43 | 48 | 142

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Time Frame: Day 0 - Day 150
Population: The safety population included all randomized subjects who received study drug and had any safety follow-up.
Measure: Number; unit: participants
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 83 | 83 | 93
participants | 19 | 7 | 11

2. Primary Outcome: Number of Subjects Reporting Adverse Events (AEs)
Time Frame: Day 0 - Day 150
Population: The safety population included all randomized subjects who received study drug and had any safety follow-up.
Measure: Number; unit: participants
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 83 | 83 | 93
participants | 77 | 75 | 83

3. Primary Outcome: Number of Subjects With Changes in Laboratory Chemistry Values Reported as AEs.
Description: Serum chemistry samples were collected at Day 0, Day 60, and Day 150. Values representing changes in severity according to the AE grading table were recorded as AEs.
Time Frame: Day 0 - Day 150
Population: The safety population included all randomized subjects who received study drug and had any safety follow-up.
Measure: Number; unit: participants
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 83 | 83 | 93
participants
  Alanine aminotransferase increased | 1 | 1 | 5
  Hepatic enzyme increased | 1 | 0 | 0
  Liver function test abnormal | 0 | 0 | 1
  Blood urea increased | 1 | 1 | 3
  Aspartate aminotransferase increased | 2 | 3 | 2

4. Secondary Outcome: The Serum Concentrations of Motavizumab at Day 0
Time Frame: Day 0
Population: The PK/immunogenicity population included all subjects in the safety population who did not receive commercial Synagis within 120 days prior to Study Day 0. Additional subjects were excluded from individual time point summaries of the analyses if the correct number of study drug doses were not received prior to the corresponding time point.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 76 | 75 | 85
μg/mL | NA (NA) — Values were below the level of detection. | NA (NA) — Values were below the level of detection. | NA (NA) — Values were below the level of detection.

5. Secondary Outcome: The Trough Serum Concentrations of Motavizumab at Day 60
Time Frame: Day 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 67 | 70 | 72
μg/mL | 74.74 (27.50) | 0.9417 (2.287) | 78.02 (28.98)

6. Secondary Outcome: The Trough Serum Concentrations of Motavizumab at Day 150
Time Frame: Day 150
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 53 | 54 | 62
μg/mL | 8.801 (5.682) | 93.05 (30.97) | 105.8 (37.49)

7. Secondary Outcome: The Trough Serum Concentrations of Motavizumab 120-150 Days Post Final Dose
Time Frame: 120-150 days post final dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 73 | 72 | 83
μg/mL | 0.5078 (1.031) | 7.586 (5.152) | 10.01 (6.341)

8. Secondary Outcome: The Serum Concentrations of Palivizumab at Day 0
Time Frame: Day 0
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 73 | 72 | 83
μg/mL | NA (NA) — Values were below the level of detection. | NA (NA) — Values were below the level of detection. | NA (NA) — Values were below the level of detection.

9. Secondary Outcome: The Trough Serum Concentrations of Palivizumab at Day 60
Time Frame: Day 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 66 | 66 | 69
μg/mL | 8.103 (6.907) | 87.37 (17.41) | 8.795 (6.578)

10. Secondary Outcome: The Trough Serum Concentrations of Palivizumab at Day 150
Time Frame: Day 150
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 52 | 54 | 60
μg/mL | 107.4 (30.21) | 22.89 (5.631) | 12.99 (7.472)

11. Secondary Outcome: The Trough Serum Concentrations of Palivizumab at 120-150 Days Post Final Dose
Time Frame: 120-150 days post final dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 72 | 71 | 81
μg/mL | 7.667 (7.719) | NA (NA) — Values were below the level of detection. | NA (NA) — Values were below the level of detection.

12. Secondary Outcome: The Immunogenicity of Motavizumab at Day 0
Description: Number of subjects with detected anti-motavivumab antibodies are reported; defined as a titer with a dilution value of greater than or equal to 1:10.
Time Frame: Day 0
Population: as for outcome 4
Measure: Number; unit: participants with detected antibody
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 77 | 80 | 89
participants with detected antibody | 0 | 1 | 0

13. Secondary Outcome: The Immunogenicity of Motavizumab at Day 60
Description: as for outcome 12
Time Frame: Day 60
Population: as for outcome 4
Measure: Number; unit: participants with detected antibody
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 76 | 82 | 90
participants with detected antibody | 0 | 0 | 0

14. Secondary Outcome: The Immunogenicity of Motavizumab at Day 150
Description: as for outcome 12
Time Frame: Day 150
Population: as for outcome 4
Measure: Number; unit: participants with detected antibody
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 73 | 75 | 84
participants with detected antibody | 1 | 1 | 0

15. Secondary Outcome: The Immunogenicity of Motavizumab at 120 to 150 Days Post Final Dose
Description: as for outcome 12
Time Frame: 120 - 150 days post final dose
Population: as for outcome 4
Measure: Number; unit: participants with detected antibody
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 75 | 74 | 84
participants with detected antibody | 3 | 1 | 0

16. Secondary Outcome: The Immunogenicity of Motavizumab at Any Time
Description: as for outcome 12
Time Frame: At any time
Population: as for outcome 4
Measure: Number; unit: participants with detected antibody
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 79 | 83 | 91
participants with detected antibody | 4 | 2 | 0

17. Secondary Outcome: The Immunogenicity of Palivizumab at Day 0
Description: Number of subjects with detected anti-palivizumab antibodies are reported; defined as a titer with a dilution value of greater than or equal to 1:10.
Time Frame: Day 0
Population: as for outcome 4
Measure: Number; unit: participants with detected antibody
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 76 | 78 | 86
participants with detected antibody | 0 | 0 | 0

18. Secondary Outcome: The Immunogenicity of Palivizumab at Day 60
Description: as for outcome 17
Time Frame: Day 60
Population: as for outcome 4
Measure: Number; unit: participants with detected antibody
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 76 | 82 | 89
participants with detected antibody | 1 | 1 | 1

19. Secondary Outcome: The Immunogenicity of Palivizumab at Day 150
Description: as for outcome 17
Time Frame: Day 150
Population: as for outcome 4
Measure: Number; unit: participants with detected antibody
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 73 | 75 | 84
participants with detected antibody | 2 | 1 | 0

20. Secondary Outcome: The Immunogenicity of Palivizumab at 120 to 150 Days Post Final Dose
Description: as for outcome 17
Time Frame: 120 - 150 days post final pose
Population: as for outcome 4
Measure: Number; unit: participants with detected antibody
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 74 | 74 | 83
participants with detected antibody | 3 | 0 | 0

21. Secondary Outcome: The Immunogenicity of Palivizumab at Any Time
Description: as for outcome 17
Time Frame: At any time
Population: as for outcome 4
Measure: Number; unit: participants with detected antibody
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Number analyzed (Participants) | 82 | 83 | 90
participants with detected antibody | 4 | 2 | 1

ADVERSE EVENTS:
Time Frame: Day 0 - Day 150
Description: Safety population
Arm/Group | Motavizumab (MEDI-524) Followed by Palivizumab | Palivizumab Followed by Motavizumab (MEDI-524) | Motavizumab (MEDI-524) Control
Serious Adverse Events (participants affected / at risk) | 19/83 | 7/83 | 11/93
Other Adverse Events (participants affected / at risk) | 75/83 | 74/83 | 83/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motavizumab (MEDI-524) Followed by Palivizumab (N=83) | Palivizumab Followed by Motavizumab (MEDI-524) (N=83) | Motavizumab (MEDI-524) Control (N=93)
Visual disturbance (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
INFANTILE COLIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
BRONCHIOLITIS (Infections and infestations) | 6 (6) | 1 (1) | 3 (3)
BRONCHITIS (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
BRONCHITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CROUP INFECTIOUS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 3 (4) | 0 (0) | 1 (1)
PNEUMONIA INFLUENZAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA PARAINFLUENZAE VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA RESPIRATORY SYNCYTIAL VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
RESPIRATORY SYNCYTIAL VIRUS BRONCHIOLIT (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
STAPHYLOCOCCAL SCALDED SKIN SYNDROME (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 0 (0) | 1 (1)
APNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motavizumab (MEDI-524) Followed by Palivizumab (N=83) | Palivizumab Followed by Motavizumab (MEDI-524) (N=83) | Motavizumab (MEDI-524) Control (N=93)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 6 (6) | 3 (3)
CONJUNCTIVITIS (Eye disorders) | 6 (6) | 11 (11) | 16 (16)
ANAEMIA NEONATAL (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 4 (4)
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 (5) | 1 (1) | 3 (3)
CONSTIPATION (Gastrointestinal disorders) | 6 (8) | 6 (6) | 6 (10)
DIARRHOEA (Gastrointestinal disorders) | 12 (13) | 13 (15) | 11 (13)
FLATULENCE (Gastrointestinal disorders) | 1 (2) | 2 (2) | 3 (5)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 4 (4) | 7 (9) | 7 (7)
INFANTILE COLIC (Gastrointestinal disorders) | 0 (0) | 1 (3) | 2 (2)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (4)
TEETHING (Gastrointestinal disorders) | 10 (24) | 9 (14) | 16 (27)
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
VOMITING (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
INJECTION SITE ERYTHEMA (General disorders) | 3 (4) | 9 (9) | 8 (13)
IRRITABILITY (General disorders) | 10 (27) | 11 (32) | 11 (43)
PYREXIA (General disorders) | 6 (6) | 8 (8) | 11 (11)
IMMUNISATION REACTION (Immune system disorders) | 3 (3) | 4 (6) | 2 (2)
BRONCHIOLITIS (Infections and infestations) | 6 (7) | 6 (6) | 2 (2)
BRONCHITIS (Infections and infestations) | 14 (21) | 20 (27) | 19 (29)
CANDIDA NAPPY RASH (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)
CANDIDIASIS (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
EAR INFECTION (Infections and infestations) | 0 (0) | 2 (3) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 7 (8) | 4 (4) | 5 (5)
GASTROENTERITIS ROTAVIRUS (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
GENITAL CANDIDIASIS (Infections and infestations) | 2 (2) | 3 (4) | 1 (1)
LARYNGITIS (Infections and infestations) | 2 (2) | 3 (4) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 (12) | 6 (8) | 6 (11)
NASOPHARYNGITIS (Infections and infestations) | 25 (35) | 26 (40) | 23 (37)
ORAL CANDIDIASIS (Infections and infestations) | 2 (3) | 5 (5) | 2 (2)
OTITIS MEDIA (Infections and infestations) | 4 (5) | 4 (4) | 4 (4)
OTITIS MEDIA ACUTE (Infections and infestations) | 2 (2) | 0 (0) | 5 (5)
PHARYNGITIS (Infections and infestations) | 7 (7) | 4 (4) | 10 (10)
RASH PUSTULAR (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
RHINITIS (Infections and infestations) | 10 (12) | 14 (18) | 8 (8)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 17 (28) | 15 (22) | 18 (25)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
VARICELLA (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
VIRAL INFECTION (Infections and infestations) | 3 (3) | 2 (2) | 3 (4)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 1 (1) | 5 (5)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 3 (3) | 2 (2)
BLOOD UREA INCREASED (Investigations) | 1 (1) | 1 (2) | 3 (3)
CARDIAC MURMUR (Investigations) | 2 (2) | 1 (1) | 2 (2)
HYPERTONIA (Nervous system disorders) | 5 (5) | 1 (1) | 0 (0)
PSYCHOMOTOR SKILLS IMPAIRED (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
AGITATION (Psychiatric disorders) | 3 (3) | 2 (3) | 2 (2)
BREATH HOLDING (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0)
GENITAL RASH (Reproductive system and breast disorders) | 1 (2) | 1 (1) | 2 (2)
BRONCHIAL HYPERREACTIVITY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 4 (5) | 5 (6)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 1 (1) | 3 (3)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 3 (12) | 5 (6) | 1 (2)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 15 (21) | 8 (11) | 10 (12)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 1 (1)
DERMATITIS DIAPER (Skin and subcutaneous tissue disorders) | 5 (5) | 10 (12) | 10 (16)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 4 (6)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (7) | 4 (7)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
RASH (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (6) | 4 (6)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.